CLINICAL TRIAL: NCT04979806
Title: A Phase 3, Randomized, Double-blind, Multicenter, Comparative Study to Determine the Efficacy and Safety of Cefepime-zidebactam vs. Meropenem in the Treatment of Complicated Urinary Tract Infection or Acute Pyelonephritis in Adults
Brief Title: Study of Cefepime-zidebactam (FEP-ZID) in Complicated Urinary Tract Infection (cUTI) or Acute Pyelonephritis (AP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wockhardt (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: W-5222-301
Record Dates: First submitted 2021-07-05; First posted 2021-07-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis
MeSH Terms: interventions — cefepime-zidebactam; Meropenem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cefepime-zidebactam (FEP-ZID) (Experimental)
  Interventions: Drug: Cefepime-zidebactam (FEP-ZID)
- Meropenem (Active Comparator)
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Cefepime-zidebactam (FEP-ZID) — 3 g (2 g FEP + 1 g ZID) IV q8h
  Arms: Cefepime-zidebactam (FEP-ZID)
Drug: Meropenem — 1 g IV q8h
  Arms: Meropenem

SUMMARY:
This is a Phase 3, randomized, double-blind, multicenter, non-inferiority study to evaluate the efficacy, safety, and tolerability of FEP-ZID vs. meropenem in the treatment of hospitalized adults with cUTI or AP.

Approximately 528 hospitalized adult subjects (≥ 18 years of age) diagnosed with cUTI or AP will be enrolled in the study. The diagnosis of cUTI or AP will be based on a combination of clinical symptoms and signs plus the presence of pyuria. The total duration of treatment with study drug is 7 to 10 days. Each subject must remain hospitalized during the study drug treatment period; no outpatient parenteral antibiotic therapy is allowed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age
2. Provide a signed written informed consent prior to any study-specific procedures
3. Meet the clinical criteria for either cUTI or AP
4. Requires hospitalization to manage the cUTI or AP
5. Agrees to use effective methods of contraception

Exclusion Criteria:

1. Known or suspected disease that may confound the assessment of efficacy.
2. Receipt of more than 72 hours of prior antibiotic therapy except for those failing prior antibiotic therapy and/or having documented uropathogen resistant to the prior therapy.
3. Rapidly progressive illness such that the subject is unlikely to survive the study period.
4. Pregnant or breastfeeding women
5. History of a seizure disorder requiring current treatment
6. Creatinine clearance < 15 mL/min or on renal dialysis
7. Neutropenia or elevated liver enzymes
8. Hypersensitivity to beta-lactam antibiotics
9. Unlikely to comply with the protocol or the Investigator considers that study participation may not be optimal for the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with overall success at Test-of-Cure | Test Of Cure Visit (Day 17 ± 2 days)
  Overall success is defined as complete resolution of cUTI or AP symptoms present at study entry (or return to premorbid state) and no new cUTI or AP symptoms together with microbiologic eradication of the bacterial pathogen found at study entry (reduced to <1000 colony forming units or CFU/mL)
Percentage of subjects with Treatment-Emergent Adverse Events (TEAE) | Day 1 to the end of study Late Follow-Up visit (LFU) (26 ± 2 days)]
  Collection of number of adverse events.

SECONDARY OUTCOMES:
Percentage of subjects with overall success at End-of-Treatment | End of Treatment Visit (Day 7 - 10 ± 1 day)
  Overall success is defined as complete resolution of cUTI or AP symptoms present at study entry (or return to premorbid state) and no new cUTI or AP symptoms together with microbiologic eradication of the bacterial pathogen found at study entry (<1000 CFU/mL)
Percentage of subjects with clinical cure at End-of-Treatment | End of Treatment Visit (Day 7 - 10 ± 1 day)
  Clinical cure is defined as complete resolution of cUTI or AP symptoms present at study entry (or return to premorbid state) and no new cUTI or AP symptoms together with microbiologic eradication of the bacterial pathogen found at study entry (reduced to <1000 CFU/mL)(CFU)/mL.
Percent of subjects with microbiological eradication at End-of-Treatment | End of Treatment Visit (Day 7 - 10 ± 1 day)
  Microbiologic eradication is defined as demonstrating <1000 CFU/mL of the bacterial pathogen found at study entry
Percentage of subjects with clinical cure at Test-of-Cure | End of Treatment Visit (Day 17 ± 2 days)
  Clinical cure is defined as complete resolution of cUTI or AP symptoms present at study entry (or return to premorbid state) and no new cUTI or AP symptoms together with microbiologic eradication of the bacterial pathogen found at study entry (reduced to <1000 CFU/mL)
Percent of subjects with microbiological eradication at Test-of-Cure | End of Treatment Visit (Day 17 ± 2 days)
  Microbiologic eradication is defined as demonstrating <1000 CFU/mL of the bacterial
Percentage of subjects with clinical cure at Late Follow-up | End of Treatment Visit (Day 26 ± 2 days)
  Clinical cure is defined as complete resolution of cUTI or AP symptoms present at study entry (or return to premorbid state) and no new cUTI or AP symptoms together with microbiologic eradication of the bacterial pathogen found at study entry (reduced to <1000 CFU/mL)
Plasma Concentration of FEP-ZID | On Days 1 and 3 of dosing prior to infusion, within 15 minutes after the end of infusion, and at 3 timepoints up to 7 hours hours post infusion

CONTACTS AND LOCATIONS:
Locations (48):
- United States (2):
  - S&D Clinical Research, LLC, Fort Myers, Florida
  - Santos Research Center, Tampa, Florida
- Bulgaria (9):
  - MHAT Dobrich AD, Dobrich
  - UMHAT Dr. Georgi Stranski, Pleven
  - Multiprofile Hospital for Active Treatment - Plovdiv AD, Plovdiv, Plovdiv
  - Multiprofile Hospital for Active Treatment - KANEV, Rousse
  - Multiprofile Hospital for Active Treatment (MHAT)- Silistra, Silistra
  - Acibadem City Clinic University Multiprofile Hospital for Active Treatment Tokuda EAD, Sofia
  - Multiprofile Hospital for Active Teatment (MHAT) and Emergency Medicine - Pirogov, Sofia
  - UMHAT Aleksandrovska Sofia - Clinic of Urology, Clinic of Anaesthesiology and Intensive Care, Clinic of Clinical Hematology, Sofia
  - Multiprofile Hospital for Active Treatment (MHAT) Sveta Anna - Varna, Varna
- China (8):
  - Hunan Provincial People's Hospital, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - Deyang People's Hospital, Deyang
  - General hospital of the PLA northern theater command, Liaoyang
  - Fudan University Huashan Hospital, Shanghai
  - Shaoxing People's Hospital, Shaoxing
- Estonia (5):
  - Ida-Viru Central Hospital, Kohtla-Järve
  - North Estonia Medical Centre Foundation, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
  - South-Estonian Hospital Ltd., Võru
- India (6):
  - Super Speciality Hospital Government Medical College and Hospital, Aurangabad, Maharashtra
  - Supe Hearth & Diabetes Hospital & Research Centre, Nashik, Maharashtra
  - ACE Hospital and Research Centre, Pune, Maharashtra
  - Accord Hospitals, Pune, Maharashtra
  - Aartham Multi Super Speciality Hospital, Ahmedabad
  - ORIION Citicare Super Speciality Hospital, Aurangabad
- Lithuania (4):
  - Klaipedos university hospital, Klaipėda
  - Republican Vilnius University hospital, Vilnius
  - Vilnius city clinical hospital, Vilnius
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Mexico (6):
  - Hospital Angeles Chihuahua, Chihuahua City
  - JM Research Cuernavaca, Cuernavaca
  - Centro de Investigacion Clinica de Oaxaca (CICLO), Oaxaca City
  - Pharmacology & Clinical Research, Querétaro
  - Arke SMO S.A. de C.V., Veracruz
  - Unidad de Atención Médica e Investigación en Salud (Unamis), Yucatán
- Poland (4):
  - Zespol Opieki Zdrowotnej w Boleslawcu, Bolesławiec
  - SCM Sp. z o.o., Krakow
  - Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego w Lodzi, Oddzial Nefrologii, Lodz
  - Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy, Klinika Chorob Wewnetrznych, Nefrologii i Dializoterapii, Warsaw
- Slovakia (4):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica, Banská Bystrica
  - Fakultna nemocnica Nitra, Nitra
  - Nemocnica Poprad, a.s. Urologicke oddeleni, Poprad
  - Fakultna nemocnica s poliklinikou Zilina, Žilina